CLINICAL TRIAL: NCT01507363
Title: Analgesic Effect of Perioperative Gabapentin in Total Knee Arthroplasty: A Randomized, Double-blind, Placebo-controlled, Dose-response Study
Brief Title: Analgesic Effect of Gabapentin in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, principal and koordinating investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THL-06-11; 2011-003105-22 (EudraCT Number); H-4-2011-082 (Registry Identifier: Ethics Committee)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Postoperative Pain; Postoperative Sedation
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gabapentin "high" (Active Comparator): Tables with Gabapentin (1300 mg/day) for 7 days, starting on the day of surgery
  Interventions: Drug: Gabapentin
- Gabapentin "intermediate" (Active Comparator): Tables with Gabapentin for 7 days (900 mg/day), starting on the day of surgery
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo tablets for 7 days, starting on the day of surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Tables with Gabapentin (1300 mg/ day) for 7 days, starting on the day of surgery
  Arms: Gabapentin "high"
Drug: Gabapentin — Tables with Gabapentin (900 mg/day) for 7 days, starting on the day of surgery
  Arms: Gabapentin "intermediate"
Drug: Placebo — Placebo tablets for 7 days, starting on the day of surgery
  Arms: Placebo

SUMMARY:
Pain is a major problem after TKA. Gabapentin may reduce acute postoperative pain. The investigators therefore investigate the effect of Gabapentin as a perioperative analgesic.

DETAILED DESCRIPTION:
Pain is a major problem after TKA. Studies indicate that Gabapentin may reduce acute postoperative pain. However, the optimal dose is unknown and there is constant controversy on analgesic versus side-effects. The investigators therefore investigate the effect of Gabapentin as a perioperative analgesic in a dose-related manner and with a sample-size allowing evaluation of side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Primary, unilateral total knee arthroplasty (TKA)
* Age 50-85 years
* Ethnic Danes

Exclusion Criteria:

* Treatment with gabapentins, systemic glucocorticoids, opioids, anxiolytic agents, antiepileptics or antidepressive agents (last 4 weeks)
* History of depression or mania
* History of alcohol or drug abuse
* History of malignancy
* History of epilepsia
* BMI > 40
* Disease affecting central or peripheral nerve function
* History of dementia
* History of renal insufficiency
* Allergy to Gabapentin
* Women with menstruation (last 2 years)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain | At 24 hour
  Pain during walking at 24 hour after surgery, visuel analog scale (VAS, 0-100 mm)

SECONDARY OUTCOMES:
Sedation | At 6 hours
  Sedation at 6 hours, numeric range scale (NRS, 0-10)
Pain | 1 week
  Pain at rest and during walking the first week after TKA, visuel analog scale (VAS, 0-100 mm)
Cumulated pain scores | 1 week
  Cumulated pain scores for pain the first week after TKA
Amount of rescue analgesic | 1 week
  Amount of rescue analgesic the first week after TKA, mg
Side effects | 1 week
  Side effects the first week after TKA
Cumulated side effects scores | 1 week
  Cumulated side effects scores the first week after TKA
Amount of ondansetron and sleeping medicine | 1 week
  Amount of ondansetron and sleeping medicine the first week after TKA, mg
Anxiety and depression | 1 week
  Anxiety and depression - questionnaire - the first week after TKA, Hospitality and Anxiety and Depression Scale
Gabapentin level in blood-sample | 1 Day
  Gabapentin level in blood-sample at 12 am on the first day after surgery, serum-koncentration

CONTACTS AND LOCATIONS:
Overall Officials: Torben B Hansen B Hansen, MD, Principal Investigator — Regionshospitalet Holstebro; Henrik Kehlet, MD, Study Director — Rigshospitalet, Denmark; Jørgen B Dahl, MD, Principal Investigator — Rigshospitalet, Denmark; Per W Kristensen, MD, Principal Investigator — Vejle Sygehus; Henrik Husted, MD, Principal Investigator — Hvidovre University Hospital; Søren Solgaard, MD, Principal Investigator — Gentofte Hospital; Mogens B Laursen, MD, Phd., Principal Investigator — Aalborg Sygehus; Lars Hansen, MD, Principal Investigator — Esbjerg Sygehus
Locations (3):
- Denmark (3):
  - Dep. of ortopedic surgery, Aalborg Sygehus, Aalborg, Aalborg
  - Dep. of ortopedic surgery, Esbjerg Sygehus, Esbjerg, Esbjerg
  - Dep. of anesthesiology and ortopedic surgery Hvidovre Hospital, Copenhagen, Hvidovre